CLINICAL TRIAL: NCT06982222
Title: A First-in-Human Dose-Finding Phase I Study of Bone-targeted High Specific Activity Stannic-117m Pentatate (Sn-117m-DTPA) in Solid Tumors With Skeletal Metastases
Brief Title: Testing the Safety of the Anti-cancer Drug, Sn-117m-DTPA, for Advanced Cancers That Have Spread to Bones
Status: Not yet recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NCI-2025-03588; NCI-2025-03588 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 10666 (Other: Ohio State University Comprehensive Cancer Center LAO); 10666 (Other: CTEP); UM1CA186712 (NIH)
Record Dates: First submitted 2025-05-20; First posted 2025-05-21 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-12

CONDITIONS: Anatomic Stage IV Breast Cancer AJCC v8; Metastatic Breast Carcinoma; Metastatic Lung Non-Small Cell Carcinoma; Metastatic Malignant Neoplasm in the Bone; Metastatic Prostate Adenocarcinoma; Stage IV Lung Cancer AJCC v8; Stage IVB Prostate Cancer AJCC v8
MeSH Terms: conditions — Breast Neoplasms; Carcinoma, Non-Small-Cell Lung; Lung Neoplasms; Prostatic Neoplasms | interventions — Specimen Handling; Magnetic Resonance Spectroscopy; Glutamate Carboxypeptidase II; X-Rays; Photons; Technetium; Pentetic Acid

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (1):
- Treatment (Sn-117m-DTPA) (Experimental): Patients receive Sn-117m-DTPA IV over 10 minutes on day 1 of each cycle. Cycles repeat every 56 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo urine and blood sample collection, PET/CT and SPECT/CT throughout the study. Additionally, prostate cancer patients undergo Tc-99m bone scan at baseline and PSMA PET/CT throughout the study.
  Interventions: Procedure: Biospecimen Collection; Procedure: Bone Scan; Procedure: Computed Tomography; Procedure: Positron Emission Tomography; Procedure: PSMA PET Scan; Procedure: Single Photon Emission Computed Tomography; Radiation: Technetium TC-99m; Radiation: Tin Sn 117m Pentetate

INTERVENTIONS:
Procedure: Biospecimen Collection — Undergo urine and blood sample collection
  Other Names: Biological Sample Collection; Biospecimen Collected; Specimen Collection
Procedure: Bone Scan — Undergo technetium TC-99m bone scan
  Other Names: Bone Scintigraphy
Procedure: Computed Tomography — Undergo PET/CT, SPECT/CT and PSMA PET/CT
  Other Names: CAT; CAT Scan; Computed Axial Tomography; Computerized Axial Tomography; Computerized axial tomography (procedure); Computerized Tomography; Computerized Tomography (CT) scan; CT; CT Scan; Diagnostic CAT Scan; Diagnostic CAT Scan Service Type; tomography
Procedure: Positron Emission Tomography — Undergo PET/CT
  Other Names: Medical Imaging, Positron Emission Tomography; PET; PET Scan; Positron emission tomography (procedure); Positron Emission Tomography Scan; Positron-Emission Tomography; PT
Procedure: PSMA PET Scan — Undergo PSMA PET/CT
  Other Names: Prostate-specific Membrane Antigen PET; PSMA PET; PSMA-Positron emission tomography
Procedure: Single Photon Emission Computed Tomography — Undergo SPECT/CT
  Other Names: Medical Imaging, Single Photon Emission Computed Tomography; Single Photon Emission Tomography; Single-Photon Emission Computed; single-photon emission computed tomography; SPECT; SPECT imaging; SPECT SCAN; SPET; ST; tomography, emission computed, single photon; Tomography, Emission-Computed, Single-Photon
Radiation: Technetium TC-99m — Undergo technetium TC-99m bone scan
  Other Names: Tc 99m; Technetium 99m
Radiation: Tin Sn 117m Pentetate — Given IV
  Other Names: PENTETATE STANNIC SN-117M; Sn 117m Pentetic Acid; Sn-117m DTPA; Tin Sn 117m DTPA

SUMMARY:
This phase I trial tests the safety, side effects and best dose of tin (Sn)-177m-diethylenetriaminepentaacetic acid (DTPA) and how well it works in treating prostate, breast or non-small cell lung cancer that has spread from where it first started (primary site) to the bones (bone metastases). Sn-117m-DTPA was originally tested in tumors that had spread to the bones to help reduce bone pain. The drug has been improved and is designed to send low-level radiation to tumors in the bone while being gentler on the bone marrow, where blood cells are made. Sn-117m-DTPA may be safe and tolerable, and may slow down or shrink tumors in patients with metastatic prostate, breast, or non-small cell lung cancer that has spread to the bones.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVE:

I. To assess the safety and tolerability of tin Sn 117m pentetate (Sn-117m- diethylenetriaminepentaacetic acid [DTPA]) per Common Terminology Criteria for Adverse Events (CTCAE), version 5.0.

SECONDARY OBJECTIVES:

I. To observe and record anti-tumor activity by prostate-specific membrane antigen (PSMA) positron emission tomography (PET) response criteria for prostate cancer and Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) response criteria for breast and non-small cell lung cancers.

II. To evaluate time to the first symptomatic skeletal event defined as (i) the first use of external-beam radiation therapy to relieve skeletal symptoms; (ii) new symptomatic pathologic vertebral or nonvertebral bone fractures; (iii) spinal cord compression; or (iv) tumor-related orthopedic surgical intervention (Scher et al., 2016).

III. To measure changes and time to progression in serum prostate-specific antigen (PSA) (in prostate cancer patients only), and bone-specific alkaline phosphatase (bALK PHOS) (in all patients).

IV. To evaluate 2-year progression-free survival (PFS) and overall survival (OS) rates.

V. To characterize the biodistribution and dosimetry of high specific activity Sn-117m-DTPA in the treated population.

OUTLINE: This is a dose-escalation study followed by a dose-expansion study.

Patients receive Sn-117m-DTPA intravenously (IV) over 10 minutes on day 1 of each cycle. Cycles repeat every 56 days for up to 4 cycles in the absence of disease progression or unacceptable toxicity. Patients also undergo urine and blood sample collection, PET/computed tomography (CT) and single photon emission computed tomography (SPECT)/CT throughout the study. Additionally, prostate cancer patients undergo technetium TC-99m (Tc-99m) bone scan at baseline and PSMA PET/CT throughout the study.

After completion of study treatment, patients are followed up every 6 months until death.

ELIGIBILITY:
Inclusion Criteria:

* Histologically documented prostate, breast, or non-small cell lung cancer (NSCLC)
* Metastatic disease in bone only (patients with visceral disease, cutaneous disease or malignant lymph nodes > 3 cm in largest diameter are not eligible)
* Documented disease progression (1 or more new bone lesion or enlargement of existing bone lesion, identified by Tc-99m bone scintigraphy or CT scan, magnetic resonance imaging [MRI], fludeoxyglucose F-18 [FDG] PET CT scan or PSMA PET CT scan)
* Must have progression on at least one line of standard of care systemic therapy. There are no maximum number of prior therapies
* Patients with prostate cancer

  * Patients with prostate adenocarcinoma, their disease must be characterized as: must have prior bilateral orchiectomy or ongoing androgen-deprivation therapy and a castrate level of serum testosterone (< 50 ng/dL or < 1.7 nmol/L)
  * Serum PSA progression, defined as two consecutive increases in PSA over a previous reference value, each measurement at least one week apart or, PSA progression ≥ 25% after 12 weeks of current standard of care (SOC) therapy (Scher et al., 2016)
  * Patients must have a baseline positive PSMA-PET scan. Patients must have progressed on at least one line of hormone therapy: Androgen receptor signaling inhibitors (ARSIs) therapy such as enzalutamide, apalutamide, darolutamide, or androgen synthesis blockers (abiraterone acetate). There are no minimum number of prior hormone therapies
  * Progression after chemotherapy (docetaxel or cabazitaxel) in patients who were chemotherapy candidates is allowed. However, prior chemotherapy is not required
  * Progression after a prostate-specific membrane antigen (PSMA)-targeted radiopharmaceutical therapy (for example: lutetium-177 vipivotide tetraxetan [Pluvicto]) is allowed but not required
  * Allowed to have received one prior cytotoxic chemotherapy treatment and one radiopharmaceutical therapy treatment OR no more than two cytotoxic chemotherapy treatments (for patients who have not received a prior radiopharmaceutical therapy treatment)
* Patients with breast cancer

  * Patients with any estrogen receptor (ER)/progesterone receptor (PR)/human epidermal growth factor receptor 2 (HER2) receptor status are eligible
  * Patients with hormone-receptor positive disease should have progressed on at least one or more prior line(s) of SOC anti-estrogen therapy and a cyclin-dependent kinase (CDK)4/6 inhibitor (except if patient had a contraindication or intolerable toxicity with the use of these agents)
  * Patients with HER2 positive disease should have progressed on at least one or more line(s) of SOC anti-HER2 therapy.
  * Patients with triple negative disease should have progressed on at least one more line(s) of SOC chemotherapy
  * Previous radiation and chemotherapy are allowed
* Patients with non-small cell lung cancer (NSCLC)

  * Patients with NSCLC should have progressed on at least one or more prior line(s) of SOC therapy, including chemotherapy and/or immunotherapy or targeted therapy if they qualify
* Age ≥ 18 years. Because no dosing or adverse event data are currently available on the use of Sn-117m-DTPA in patients < 18 years of age, children are excluded from this study
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2 (Karnofsky ≥ 60%)
* Absolute neutrophil count ≥ 1,000/mcL
* Platelets ≥ 75,000/mcL
* Hemoglobin > 9 g/dL
* Total bilirubin ≤ 2.5 x institutional upper limit of normal (ULN)
* Aspartate aminotransferase (AST)(serum glutamic oxaloacetic transaminase [SGOT])/alanine aminotransferase (ALT)(serum glutamic pyruvic transaminase [SGPT]) ≤ 5 x institutional ULN
* Creatinine ≤ 1.7 mg/dL OR glomerular filtration rate (GFR) ≥ 50 mL/min/1.73 m^2
* Patients must be taking a bone health agent (bisphosphonates or denosumab) for at least one (1) month prior to enrollment
* Human immunodeficiency virus (HIV)-infected patients on effective anti-retroviral therapy with undetectable viral load within 6 months are eligible for this trial
* For patients with evidence of chronic hepatitis B virus (HBV) infection, the HBV viral load must be undetectable on suppressive therapy, if indicated
* Patients with a history of hepatitis C virus (HCV) infection must have been treated and cured. For patients with HCV infection who are currently on treatment, they are eligible if they have an undetectable HCV viral load
* Patients with treated brain metastases are eligible if follow-up brain imaging after central nervous system (CNS)-directed therapy shows no evidence of progression
* Patients with a prior or concurrent malignancy whose natural history or treatment does not have the potential to interfere with the safety or efficacy assessment of the investigational regimen are eligible for this trial
* Patients with known history or current symptoms of cardiac disease, or history of treatment with cardiotoxic agents, should have a clinical risk assessment of cardiac function using the New York Heart Association Functional Classification. To be eligible for this trial, patients should be class II or better
* The effects of Sn-117m-DTPA on the developing human fetus are unknown. For this reason and because radionucleotides are known to be teratogenic, male participants and their female partners of childbearing potential must agree to use adequate contraception (hormonal or barrier method of birth control; abstinence) prior to study entry and for the duration of study participation. A woman of childbearing potential is a premenopausal female capable of becoming pregnant. Should a woman of childbearing potential become pregnant or suspect she is pregnant while her male partner is participating in this study, she should inform her treating physician immediately. Both men and women of childbearing potential treated or enrolled on this protocol must also agree to use adequate contraception prior to the study, for the duration of study participation, and for 6 months after completion of Sn-117m-DTPA administration. For prostate cancer patients, androgen deprivation therapy is considered adequate contraception
* Ability to understand and the willingness to sign a written informed consent document. Legally authorized representatives may sign if the patient is physically (not mentally) not capable of signing

Exclusion Criteria:

* Patients who have not recovered from reversible adverse events due to prior anti-cancer therapy (i.e., have residual toxicities > grade 1) with the exception of alopecia
* Patients must not have received any investigational agents within 4 weeks or 5 half-lives, whichever is shorter, before starting study treatment, nor be scheduled to receive one during the planned treatment period
* Patients must not have a history of allergic reactions attributed to compounds of similar chemical or biologic composition to Sn-117m-DTPA
* Patients must not have imminent or established spinal cord compression, pathological fracture in weight bearing bones, or bone lesion with soft tissue component unless treated as appropriate with radiation and/or surgery before starting on this study
* Patients must not have received prior systemic radiotherapy with strontium-89, samarium-153, rhenium-186, rhenium-188, or radium-223 dichloride (Xofigo) for the treatment of bony metastases. Prior systemic radiopharmaceutical therapy with lutetium Lu 177 vipivotide tetraxetan (Pluvicto) is permitted, but last treatment must be at least six weeks prior to starting study treatment due to the concern of bone marrow suppression
* Patients must not have unmanageable urinary incontinence
* Pregnant women are excluded from this study because Sn-117m-DTPA is a radionucleotide with the potential for teratogenic or abortifacient effects. Because there is an unknown but potential risk for adverse events in nursing infants secondary to treatment of the mother with Sn-117m-DTPA, breastfeeding should be discontinued if the mother is treated with Sn-117m-DTPA

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 24 (Estimated)
Dates: Start 2026-03-31 (Estimated); Primary Completion 2027-02-12 (Estimated); Study Completion 2027-02-12 (Estimated)

PRIMARY OUTCOMES:
Frequency of dose-limiting toxicities | Up to completion of 1 cycle (cycle length = 56 days)
  Will be graded using National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) version (v) 5.0. Will be summarized by severity grade, system organ class, and their relation to study treatment.
Frequency of adverse events | Up to 30 days after last dose of study treatment
  Will be graded using NCI CTCAE v 5.0. Will be summarized by severity grade, system organ class, and their relation to study treatment.

SECONDARY OUTCOMES:
Tumor response | Up to 2 years
  Will be evaluated using prostate-specific membrane antigen (PSMA) positron emission tomography (PET)/computed tomography (CT) for prostate cancer and Positron Emission Tomography Response Criteria in Solid Tumors (PERCIST) for breast and non-small cell lung cancers. Categorical endpoints will be summarized by frequency and percent. Continuous variables will be summarized by mean and standard deviation at each assessment time point.
Time to first symptomatic skeletal event | Up to 2 years
  Will be defined as the first use of external-beam radiation therapy to relieve skeletal symptoms, new symptomatic pathologic vertebral or non-vertebral bone fractures, spinal cord compression or tumor-related orthopedic surgical intervention. Categorical endpoints will be summarized by frequency and percent. Continuous variables will be summarized by mean and standard deviation at each assessment time point. Will be analyzed using the Kaplan-Meier product limit method. Estimation and confidence intervals for the median time to first symptomatic skeletal event will be provided.
Changes in serum PSA (prostate cancer patients only) | At baseline, days 44-56 of cycle 1, and days 30-56 of cycle 2
  Categorical endpoints will be summarized by frequency and percent. Continuous variables will be summarized by mean and standard deviation at each assessment time point. Will be calculated for each of the above defined categories with the corresponding confidence intervals.
Time to progression in serum PSA (prostate cancer patients only) | At baseline, days 44-56 of cycle 1, and days 30-56 of cycle 2
  Categorical endpoints will be summarized by frequency and percent. Continuous variables will be summarized by mean and standard deviation at each assessment time point. Will be calculated for each of the above defined categories with the corresponding confidence intervals.
Changes in bone-specific alkaline phosphatase levels (all patients) | At baseline, days 44-56 of cycle 1, and days 30-56 of cycle 2
  Categorical endpoints will be summarized by frequency and percent. Continuous variables will be summarized by mean and standard deviation at each assessment time point. Will be calculated for each of the above defined categories with the corresponding confidence intervals.
Progression-free survival | From the first study treatment until the date of PERCIST definition of progression for breast and non-small cell lung cancers and PSMA PET/CT definition of progression for prostate cancer, assessed up to 2 years
  Categorical endpoints will be summarized by frequency and percent. Continuous variables will be summarized by mean and standard deviation at each assessment time point. Will be analyzed using the Kaplan-Meier product limit method.
Overall survival | From the first study treatment until the date of death, assessed up to 2 years
  Categorical endpoints will be summarized by frequency and percent. Continuous variables will be summarized by mean and standard deviation at each assessment time point. Will be analyzed using the Kaplan-Meier product limit method.
Biodistribution and dosimetry of high specific activity tin (Sn)-117m-diethylenetriaminepentaacetic acid (DTPA) | On days 1, 2, 4, and 43 of cycle 1
  Categorical endpoints will be summarized by frequency and percent. Continuous variables will be summarized by mean and standard deviation at each assessment time point. All results are expressed as mean percent of injected dose +/- standard deviation; the mean values will be tested by Student t test for statistical significance. Regions of interest will be drawn over normal bone and metastatic foci, and decay-corrected counts of pixels drawn from all Sn-117m-DTPA scans. Counts per pixels will be plotted against time. Time to peak was noted for both normal and metastatic bone lesions. The slope of the curve will be assessed for evidence of washout.

CONTACTS AND LOCATIONS:
Overall Officials: Zin W Myint, Principal Investigator — Ohio State University Comprehensive Cancer Center LAO

IPD SHARING:
Plan to Share IPD: Yes
NCI is committed to sharing data in accordance with NIH policy. For more details on how clinical trial data is shared, access the link to the NIH data sharing policy page.
URL: https://grants.nih.gov/policy/sharing.htm